CLINICAL TRIAL: NCT06834984
Title: Ritual Synbiotic+, a Dietary Supplement
Brief Title: Ritual Synbiotic+, a Dietary Supplement Designed to Impact Gastrointestinal Health, Mood, and Behavior in Women
Acronym: SYN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Ritual (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 6393
Record Dates: First submitted 2025-02-03; First posted 2025-02-19 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Gastrointestinal Disease Symptoms
Keywords: Women with gastrointestinal symptoms; Probiotic; Prebiotic
MeSH Terms: interventions — Prebiotics; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Some of the sponsor staff will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (probiotic supplement) (Experimental): This group will take a once daily supplement containing pre-pro-post biotics.
  Interventions: Dietary Supplement: Prebiotic, probiotic, postbiotic combination
- Control (Placebo Comparator): This group will be taking a once daily placebo pill.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic, probiotic, postbiotic combination — The product consists of two probiotics, Lactobacillus rhamnosus LGG and Bifidibacterium animalis subsp. lactis BB-12, supplied at a total concentration of 11B CFU's, a prebiotic consisting of 1 × 106 Plaque Forming Units (PFU) LH01-Myoviridae, LL5-Siphoviridae, T4D-Myoviridae, and LL12-Myoviridae bacteriophages, marketed as PreforPro, and tributyrin- a stale form of butyrate
  Arms: Treatment Group (probiotic supplement)
Dietary Supplement: Placebo — Placebo pill containing stomach acid-resistant outer vegan capsule (hypromellose, gellan gum), hi oleic safflower oil, inner vegan capsule (hypromellose, gellan gum) microcrystalline cellulose, ascorbyl palmitate, silica
  Arms: Control

SUMMARY:
The aim of this study is to determine how regular consumption of Synbiotic+, a dietary supplement that contains prebiotics, probiotics, and postbiotics, impacts functional gastrointestinal health, markers of intestinal inflammation and immune health, and influences mood and behavior. The primary outcome will be to assess gastrointestinal health using bowel movement tracking, self-report and objective assessments of gastrointestinal symptom severity, stool levels of short chain fatty acids, changes in the gut microbiota, including recovery of LGG and BB-12, and functional measures of the microbiome. Secondary outcomes will include stool and blood markers of gut barrier function and intestinal inflammation, immune health, and self-assessments of stress, anxiety, sleep, and quality of life.

DETAILED DESCRIPTION:
The trial will be a double-blinded, randomized, placebo-controlled parallel arm intervention study taking place at Colorado State University. In total, ~100 adult women (25-65 years old) with a BMI <30, with moderate digestive discomfort (as evidenced by a moderate score on a functional gastrointestinal questionnaire will be enrolled into the study. With an estimated 20% attrition rate, this will allow approximately 80 individuals to complete the study. Exclusion criteria include a BMI>30, any significant systemic diseases (including Crohn's, Ulcerative Colitis, but not including diagnosis of Irritable Bowel Syndrome), prescription medication for digestive symptoms, antibiotic or probiotic ingestion within the two months before entry into the study, and pregnancy or breastfeeding. Subjects will be provided with the consent form prior to the baseline visit and informed consent will be obtained prior to participating in the study. Participants will be compensated for their participation. Medical health history will be collected at the baseline visit. Quality of Life (QOL) and GI Health questionnaires, along with questionnaires to gauge mood and anxiety, will be collected from each enrolled participant at the baseline, mid-point ("check-in visit 2"), and final clinic visits; a GI health questionnaire will also be collected at the acute study visit (48-72 hours after treatment start). Anthropometric measures at the baseline visit will include seated blood pressure, height, weight, and waist:hip measurements; blood pressure will also be collected at the final visit. A stool sample will be collected from participants at each clinic visit, and a blood sample will be collected at the baseline and final clinical visits. Two 3-day diet records will be completed prior to the start and at completion of the study. In addition, participants will keep a daily record of their bowel movements and brief notes regarding any GI symptoms starting 7-days prior to beginning the treatment and for the duration of the study.

All enrolled participants will start with a baseline clinic visit and a 7-day lead in period, after which they will take one of the treatments for 12 weeks. To determine the acute effects of the treatment, participants will return a stool sample to the clinic 48-72 hours after the treatment start to establish acute effects (ie. changes in SCFA, microbial dysbiosis index). Subjects will randomly be assigned to a starting treatment (A or B) and capsules will be blinded and labeled by Ritual personnel who are not directly involved in the study. CSU clinical personnel will not be provided with the code for treatment groups until after all data analysis has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult women (age 25-65, with target average age of 50).
* BMI <30.
* with moderate gastrointestinal symptoms.
* Participants should be willing to follow the study protocol and attend clinic visits.

Exclusion Criteria:

* less than 25 years of age or greater than 65 years of age.
* have a BMI >30.
* taken antibiotics within two months or any probiotic supplements within the past 14 days prior to the start of treatment.
* current medications and dietary supplements will be assessed on a case-by- case basis and will result in exclusion if there is the possibility that the drugs or supplements used would influence the endpoints of the study. This would include statins, metformin, NSAIDs, MAO inhibitors, and hormone therapies.
* Individuals with current disease diagnosis, including diagnosis of cancer, liver or kidney disease, gastrointestinal diseases, and cardiometabolic disorders (cardiovascular disease, diabetes, etc.)
* pregnant and breastfeeding people.
* overuse of alcohol as determined on a case-by-case self-reported alcohol use.
* if the individual feels they are unable to adhere to the study requirements, which includes consuming capsules, providing stool or blood samples, tracking bowel movements and symptoms, and attending scheduled clinic visits.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Short Chain Fatty Acid concentration in stool | 4X: baseline, acute (3 days), mid-point (6 weeks), final (12 weeks).
  Gas chromatography will be used to measure changes in SCFA production in stool.
Fecal pH | 4X: baseline, acute (3 days), mid-point (6 weeks), final (12 weeks).
  Stool sample pH will be measured before and after treatment.
Fermentation Rate of microbiome | 4X: baseline, acute (3 days), mid-point (6 weeks), final (12 weeks).
  This is a functional measure of the microbiome and will be measured ex-vivo Radio Frequency Identification (RFID) system. Stool sample microbes will be assessed for fermentation rates.
Microbial composition (alpha and beta diversity, dysbiosis index, differential taxa) | 2X: baseline, and final (12 weeks)
  Changes in microbiota profiles, ratio of pro-inflammatory to beneficial microbes, recovery of LGG & BB-12 in stool; measured using 16s rRNA and targeted assays.
Total number and types of bowel movements | Daily for 12 weeks
  Defecation frequency and proportion of abnormal to normal bowel movements as recorded in a diary using the Bristol Stool Form Scale. The scale runs from 1-7 with healthier outcomes associated with 3-5 on the Bristol scale.
Gastrointestinal Symptom Rating Scale | 4X: baseline, acute (3 days), mid-point (6 weeks), final (12 weeks).
  Measures Abdominal Pain Heartburn Acid Regurgitation Sucking Sensations in the Epigastrium Nausea & Vomiting Borborygmus (rumbling) Abdominal Distension (bloating) Eructation (burping) Flatus (gas) Decreased or Increased Passage of Stools Loose or Hard Stools Urgent Need for Defecation Feeling of Incomplete Evacuation Rated on a scale starting at "No Discomfort at all" to "Very severe discomfort", where better outcomes are associated with "No Discomfort At All" while worse outcomes are associated near(er) to "Very Severe Discomfort".

SECONDARY OUTCOMES:
Fecal calprotectin | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  Intestinal inflammation
Alpha-1 antitrypsin | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  Gut permeability
Lipopolysaccharide binding protein and soluble CD14 in blood | 2X: baseline, and final (12 weeks)
  Barrier function: Lipopolysaccharide binding protein and soluble CD14 are involved in binding LPS and initiating systemic inflammatory cascades and have been used as a proxy for gut barrier function.
Human high sensitivity T-cell panel/Peripheral blood mononuclear cells (PBMCs) | 2X: baseline, and final (12 weeks)
  Immune health: in supernatants from LPS-stimulated PBMC; uses Milliplex MAP
Alpha-1 antitrypsin in blood | 2X: baseline, and final (12 weeks)
  Gut permeability/malabsorption
Cortisol blood levels | 2X: baseline, and final (12 weeks)
  Cortisol levels
GLP-1 | 2X: baseline, and final (12 weeks)
  GLP-1 levels, metabolic health, measured with ELISA assay.
Quality of Life as measured by Inflammatory Bowel Disease (IBD) Specific Quality of Life survey | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  Online Survey measuring Helplessness, Embarrassment, Vulnerability, Discomfort, Enjoyment of Life, Body Image, Depression, Isolation, Behavior Change, Anger, and Irritability in regards to bowel problems.
  Survey scale starts at "not at all" and goes up to "extremely" with healthier outcomes associated with "not at all".
Generalized Anxiety Disorder 7 Item Survey | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  The GAD-7 (Generalized Anxiety Disorder-7) is a self-report questionnaire designed to screen for generalized anxiety disorder (GAD) and assess the severity of anxiety symptoms in individuals. It consists of 7 questions that focus on the frequency of anxiety-related symptoms experienced over the past two weeks.
  Scoring:
  0-4: Minimal or no anxiety 5-9: Mild anxiety 10-14: Moderate anxiety 15-21: Severe anxiety
Positive and Negative Affect Schedule | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  Subjective experience of mood (how you feel on average) rated on a scale from "very slightly or none at all" to "extremely". Moods can be positive (e.g inspiration) or negative (e.g. guilty), so the score does not reflect a better or worse outcome.
Perceived Stress Scale | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  Subjective experiences of stress. The questions in this scale ask about your feelings and thoughts during the last month. In each case, you will be asked to indicate how often you felt or thought a certain way. The scale ranges from "never" to "very often". Questions are regarding positive and negative situations, so a total score is not indicative of a better or worse outcome.
Ritual Marketing Interest measuring the user experience of the probiotic supplement. | 3X: baseline, mid-point (6 weeks), final (12 weeks)
  Subjective experiences regarding smell, taste, ingestion, tolerability, nausea, burping, after taking the product. Also asks whether the participant would recommend the product, enjoyed the overall experience, easy to incorporate into daily routine, whether it improved skin and/or stomach discomfort.
  The survey uses a Likert Scale for all questions. Each question is situational in that the lower score, "Strongly Disagree" or the higher score "Strongly Agree" do not correlate as a "better" or "worse" outcome across all questions.
Blood Glucose levels | 2X: baseline, final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Alanine Aminotransferase (ALT) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Aspartate Aminotransferase (AST) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Alkaline Phosphatase (ALP) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Blood Creatinine | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Blood bilirubin | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Total Cholesterol | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
High Density Lipoprotein (HDL) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Blood Triglycerides | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Non-HDL Cholesterol (nHDLc) | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Total Cholesterol to HDL ratio (TC/H) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Low Density Lipoprotein (LDL) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.
Very low density lipoprotein (VLDL) in blood | 2X: baseline, and final (12 weeks)
  Measured with a point of care instrument (Piccolo Express) using a disc-based photometric analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University Food and Nutrition Clinical Research Laboratory, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No